CLINICAL TRIAL: NCT00074841
Title: A Phase II/III, Randomized, Comparative Trial of Azithromycin Plus Chloroquine Versus Sulfadoxine-Pyrimethamine Plus Chloroquine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in India
Brief Title: Trial of Azithromycin Plus Chloroquine Versus Sulfadoxine-Pyrimethamine Plus Chloroquine for the Treatment of Uncomplicated Malaria in India
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Purpose: Treatment
Other Study IDs: A0661120
Record Dates: First submitted 2003-12-22; First posted 2003-12-24 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: PLASMODIUM FALCIPARUM MALARIA
Keywords: MALARIA; INDIA; CHLOROQUINE; PLASMODIUM FALCIPARUM; SULFADOXINE-PYRIMETHAMINE
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Azithromycin; Chloroquine; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Azithromycin/Chloroquine
Drug: Sulfadoxine-Pyrimethamine/Chloroquine

SUMMARY:
This primary objective of this study is to assess whether the combination of Azithromycin with chloroquine is non-inferior to the combination of sulfadoxine-pyrimethamine plus chloroquine, when used to treat uncomplicated cases of malaria due to Plasmodium falciparum in adults in India.

ELIGIBILITY:
INCLUSION CRITERIA:

* Females and males >=18 years of age with uncomplicated, symptomatic malaria as indicated by the presence of both of the following: a.) Blood smears positive for Plasmodium falciparum asexual parasitemia between 1000 -100,000 parasites/uL; b.) Fever or history of fever ( >=38.5C/101.2F rectal or tympanic; >=37.5C/99.5F axillary or >=38C/100.4F oral) within the prior 24 hours
* Serum glucose >= 60 mg/dL (by fingerstick or peripheral blood collection)
* Positive rapid diagnostic test (Binax NOW ICT) positive for P. falciparum
* Women of childbearing potential must have a negative urine gonadotropin prior to entry into the study and must agree to use adequate contraception during the entire study

EXCLUSION CRITERIA:

* Severe or complicated malaria including subjects with any of the following: a.) Impaired consciousness (e.g. obtundation, unarousable coma), seizures or abnormal neurologic exam suggestive of severe or complicated malaria; b.) Hemoglobinuria; c.) Jaundice; d.) Respiratory distress (respiratory rate >=30/min); e.) Persistent vomiting; f.) Hematuria, as reported by the patient
* Pregnant or breast-feeding women
* History of allergy to or hypersensitivity to azithromycin or any macrolide, sulfonamides, pyrimethamine, or chloroquine
* Known or suspected folate deficiency
* Known history of blood dyscrasias (e.g., megaloblastic anemia, agranulocytosis, aplastic anemia, thrombocytopenia, leukopenia, neutropenia, hemolytic anemia)
* Known G-6PD deficiency
* History of epilepsy or psoriasis
* History of treatment with any antimalarial drug (chloroquine, quinine, mefloquine, Malarone, SP, artemisinin compounds) or antibacterial with known antimalarial activity (macrolides, doxycycline, clindamycin) within 2 weeks prior to enrollment into the study
* Known or suspected cardiovascular, hepatic or renal abnormality that in the opinion of the Investigator would place the subject at increased risk to participate in the study. The following findings are specific exclusions: a.) Serum creatinine >2.0 x ULN; b.) ALT and/or AST >3 x ULN
* Inability to swallow oral medication in tablet form
* Treatment with other investigational drugs within 30 days prior to enrollment into the study
* Alcohol and/or any other drug abuse
* Requirement to use medication during the study that might interfere with the evaluation of the study drug
* Specific systemic diseases or other medical conditions that would interfere with the evaluation of the therapeutic response or safety of the study drug
* Inability to comprehend and/or unwillingness to follow the study protocol
* Prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2003-09; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Pfizer Investigational Site, Dispur Guwahati, Assam
  - Pfizer Investigational Site, Bambolim, Gao
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Parel Mumbai, Maharashtra
  - Pfizer Investigational Site, Rourkela, Odisha
  - Pfizer Investigational Site, Vellore, Tamil Nadu
  - Pfizer Investigational Site, Indore